CLINICAL TRIAL: NCT00340613
Title: A School Intervention: Lunch Time Insulin Injections in Children With Poorly Controlled Type 1 Diabetes
Brief Title: Lunch Time Insulin Injection by School Nurse for Poorly Controlled Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Sponsored Programs, Principal Investigator, Baylor College of Medicine
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-16630
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2016-07-14 (Estimated); Status verified 2016-07

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 Diabetes; Poorly controlled glucose; adolescents
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: glargine insulin

SUMMARY:
We hypothesize that checking blood sugar and taking long and short acting insulin before lunch at school may improve overall blood sugar control, grades, and decreases school absences in children and teens with poorly controlled T1DM.

DETAILED DESCRIPTION:
The Diabetes Control and Complications Trial (DCCT), for type 1Diabetes (T1DM), showed the importance of intensified diabetes control in helping reduce complications associated with poorly controlled diabetes. However, adolescents with T1DM continue to be a high-risk population due to the difficulties in coping with the physical, emotional, and social demands associated with managing diabetes themselves.

We propose to use the school nurse to help with lunchtime blood sugar monitoring (BSM) and with a lunchtime insulin injection. We want to see if this will improve blood sugar control, improve school grades, and decrease absences from school in adolescents with poorly controlled diabetes. Subjects will receive 12 weeks of this treatment to see if they will have improved glucose control. We hope to improve blood sugar control, school grades and decrease absences from school in teens with poorly controlled diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Child with T1DM for at least 1 year
* Age 10-19 years
* Have a Hgb A1C greater than or equal to 9.0% but less than or equal 13.9% for at least 6 months.
* School must have a school nurse

Exclusion Criteria:

* Child who has Type 2 diabetes
* Subject receiving home schooling

Ages: 10 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 36 (Actual)
Dates: Start 2006-06; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Hemoglobin A1c | At the start of the study and again in 3 months

SECONDARY OUTCOMES:
Urine microalbumin | At the beginning and the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Rubina A Heptulla, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Texas Children's Diabetes Center, Houston, Texas, United States

REFERENCES:
- [Derived] Nguyen TM, Mason KJ, Sanders CG, Yazdani P, Heptulla RA. Targeting blood glucose management in school improves glycemic control in children with poorly controlled type 1 diabetes mellitus. J Pediatr. 2008 Oct;153(4):575-8. doi: 10.1016/j.jpeds.2008.04.066. PMID 18847622